CLINICAL TRIAL: NCT03165968
Title: Test and Evaluation of Non-Invasive Neuro-Assessment Devices (NINAD): NeuroKinetics, Inc, iPAS
Acronym: NINADiPAS
Status: Suspended | Type: Observational
Why Stopped: COVID19 epidemic, and institutional guidelines for halt of recruitment during epidemic
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Rapp, Director, Traumatic Injury Research Program, Uniformed Services University of the Health Sciences
Other Study IDs: MEM 91-2714
Record Dates: First submitted 2017-05-09; First posted 2017-05-24 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Neuro Kinetics, Inc, i-PAS — This is a test of i-PAS device reliability only.

SUMMARY:
The long term goal for the Traumatic Injury Research Program (TIRP) is testing of novel devices for the identification and longitudinal assessment of traumatic brain injury (TBI). The Department of Defense (DoD) has now tasked TIRP with the test and evaluation of these devices to assess reliability and validity. The objective of this effort is to test the reliability of the NeuroKinetics Inc (NKI), i-PAS (portable assessment system) device using a test/re-test protocol with healthy controls.

The basic research design adopted here is the test/re-test paradigm with three assessments obtained on three separate visits. This will allow the assessment of reliability of both the device and the measure(s) that are computed from the input signals. Participants will be Healthy Controls (HC) as defined in the inclusion exclusion section.

In this initial study we will be administering standardized self-report instruments ( Short Form - 36 (SF-36) and the Symptom Checklist-90 (SCL-90r)), standard three-lead electrocardiogram. In addition we will administer the NKI i-PAS specific protocol as delineated by NKI.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 18 and 55 years old in good general health. Good general health is operationalized for the purpose of this study by scores within one standard deviation of the mean in all eight sections of the Short Form 36 (SF-36).

A normalized Global Severity Scale of less than or equal to 65 on the Symptom Checklist-90-Revised and subscale scores less than the cut scores indicating significant pathology.

Exclusion Criteria:

* A TBI positive event as determined by the DVBIC (Defense and Veterans Brain Injury Center) Three Question Screening Tool.

Any history of seizures or CNS tumors

A normalized Global Severity Scale of more than 65 on the Symptom Checklist-90-Revised. Any subscale score indicating significant pathology

Scores greater than one standard deviation from the mean on all eight sections of the Short Form 36 (SF-36)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy control population
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Reliability of NKI i-PAS signals across three separate visits | Three measures over Four weeks (First visit; Second visit 2-6 days later; Third visit 4 weeks after first visit
  The NKI i-PAS device should provide similar signals each time a healthy control participant is tested.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - The Citadel - Military College of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Upload to FITBIR Database NIH